CLINICAL TRIAL: NCT04509609
Title: Clinical Determinants of Disease Progression in Patients With Limb Girdle Muscular Distrophy Type 2E
Acronym: NeuroLGMD2E
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 000000
Record Dates: First submitted 2020-07-09; First posted 2020-08-12 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: LGMD2E
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2E

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMD 2E with a genetic diagnosis: Any patient affected by LGMD 2E with a genetic diagnosis
  Interventions: Other: Exon 3 truncating mutation; Other: Any other mutation in SGBC gene

INTERVENTIONS:
Other: Exon 3 truncating mutation — Any patient affected by LGMD 2E with a genetic diagnosis carrying the truncating mutation c.377_384duplCAGTAGGA on exon 3, both in homozygosis and in heterozygosis
Other: Any other mutation in SGBC gene — Any patient affected by LGMD 2E with a genetic diagnosis other than the truncating mutation c.377_384duplCAGTAGGA on exon 3, both in homozygosis and in heterozygosis

SUMMARY:
A retrospective observational study that will enable us to collect retrospective data from the clinical records of LGMD 2E patients in order to highlight any possible correlation between:

* clinical variables and patient age,
* clinical variables and other clinical variables,
* clinical variables and clinical outcomes. The study will help to define the natural history of this rare disease and to ameliorate the management of these patients.

DETAILED DESCRIPTION:
Retrospective observational study. Retrospective data from clinical charts of patients affected by LGMD 2E will be collected after the subscription of informed consent.Data considered will include any clinical variable measured, both objective and subjective. All data obtained will be anonimized before any treatment. Data will be grouped according to the age of the patient, in order to have more data for each age and to gain a trustable description of the disease progression. The possible correlation of each variable to age, to other variables and to objective clinical outcomes will be studied. Clinical outcomes considered will include age of loss of deambulation, age of introduction of respiratory assist, age of introduction of cardiological therapy. Data collected will also be divided in two groups according to different genetic diagnosis in order to evaluate phenotipical differences of genotypical clesses. First group will count all patient with the truncating mutation c.377_384duplCAGTAGGA in exon 3, both in heterozigosis and in homozigosis Second group will include all the other patients.

Both on the global data collection and on data divided according to genotype, statistical analysis will be performed. Those analysis will study linear regression both with the univariate, bivariate and multivariate model.

ELIGIBILITY:
Inclusion Criteria:

* Gene based diagnosis of LGMD 2E
* Subscription of informed consent when applicable

Exclusion Criteria:

* Lacking gene based diagnosis of LGMD 2E
* Lacking subscription of informed consent when applicable

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient affected by LGMD 2E that have received a genetical confirm of the diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Natural history | december 2020
  The clinical progression of the disease will be studied considering for each clinical variable its evolution according to patients' ages. This both in overall cohort and in genetic subgroups.

SECONDARY OUTCOMES:
Guidelines | december 2020
  The collection of clinical variables describing the progression of the disease will enable a better clinical management of these patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided
under EU GDPR, this would be extremely complex

DOCUMENTS (2):
  • Study Protocol (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04509609/Prot_000.pdf
  • Informed Consent Form (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04509609/ICF_001.pdf